CLINICAL TRIAL: NCT00659425
Title: A Phase 1, Multicenter, Dose Escalation Study of CAT-8015 in Children, Adolescents and Young Adults With Refractory CD22+ Acute Lymphoblastic Leukemia (ALL) or Non-Hodgkin Lymphoma (NHL)
Brief Title: CAT-8015 in Children, Adolescents and Young Adults With Acute Lymphoblastic Leukemia or Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAT-8015-1004
Record Dates: First submitted 2008-04-10; First posted 2008-04-16 (Estimated); Results first posted 2017-10-02 (Actual); Last update posted 2017-10-02 (Actual); Status verified 2017-08

CONDITIONS: Acute Lymphoblastic Leukemia; Non-Hodgkin's Lymphoma
Keywords: Moxetumomab pasudotox
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Non-Hodgkin | interventions — immunotoxin HA22

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (10):
- 5 microgram per kilogram (mcg/kg) (Experimental): Participants received intravenous infusion of 5 mcg/kg moxetumomab pasudotox (CAT-8015) without concomitant corticosteroid administration every other day (QoD) in a 21-day cycle for a total of 6 doses per cycle.
  Interventions: Drug: CAT-8015 (Moxetumomab Pasudotox)
- 10 microgram per kilogram (mcg/kg) (Experimental): Participants received intravenous infusion of 10 mcg/kg moxetumomab pasudotox (CAT-8015) without concomitant corticosteroid administration every other day (QoD) in a 21-day cycle for a total of 6 doses per cycle.
  Interventions: Drug: CAT-8015 (Moxetumomab Pasudotox)
- 20 microgram per kilogram (mcg/kg): Schema A (Experimental): Participants received intravenous infusion of 20 mcg/kg moxetumomab pasudotox (CAT-8015) without concomitant corticosteroid administration every other day (QoD) in a 21-day cycle for a total of 6 doses per cycle.
  Interventions: Drug: CAT-8015 (Moxetumomab Pasudotox)
- 20 microgram per kilogram (mcg/kg): Schema B (Experimental): Participants received intravenous infusion of 20 mcg/kg moxetumomab pasudotox (CAT-8015) with concomitant corticosteroid administration every other day (QoD) in a 21-day cycle for a total of 6 doses per cycle.
  Interventions: Drug: CAT-8015 (Moxetumomab Pasudotox)
- 30 microgram per kilogram (mcg/kg): Schema A (Experimental): Participants received intravenous infusion of 30 mcg/kg moxetumomab pasudotox (CAT-8015) without concomitant corticosteroid administration every other day (QoD) in a 21-day cycle for a total of 6 doses per cycle.
  Interventions: Drug: CAT-8015 (Moxetumomab Pasudotox)
- 30 microgram per kilogram (mcg/kg): Schema B (Experimental): Participants received intravenous infusion of 30 mcg/kg moxetumomab pasudotox (CAT-8015) with concomitant corticosteroid administration every other day (QoD) in a 21-day cycle for a total of 6 doses per cycle.
  Interventions: Drug: CAT-8015 (Moxetumomab Pasudotox)
- 40 microgram per kilogram (mcg/kg): Schema B (Experimental): Participants received intravenous infusion of 40 mcg/kg moxetumomab pasudotox (CAT-8015) with concomitant corticosteroid administration every other day (QoD) in a 21-day cycle for a total of 6 doses per cycle.
  Interventions: Drug: CAT-8015 (Moxetumomab Pasudotox)
- 32 microgram per kilogram (mcg/kg): Schema C (Experimental): Participants received intravenous infusion of 32 mcg/kg moxetumomab pasudotox (CAT-8015) of process 3 material every other day (QoD) in a 21-day cycle for a total of 10 doses per cycle.
  Interventions: Drug: CAT-8015 (Moxetumomab Pasudotox)
- 50 microgram per kilogram (mcg/kg): Schema B (Experimental): Participants received intravenous infusion of 50 mcg/kg moxetumomab pasudotox (CAT-8015) without concomitant corticosteroid administration every other day (QoD) in a 21-day cycle for a total of 6 doses per cycle.
  Interventions: Drug: CAT-8015 (Moxetumomab Pasudotox)
- 50 microgram per kilogram (mcg/kg): Schema C (Experimental): Participants received intravenous infusion of 50 mcg/kg moxetumomab pasudotox (CAT-8015) continuous every other day (QoD) in a 21-day cycle for a total of 10 doses per cycle.
  Interventions: Drug: CAT-8015 (Moxetumomab Pasudotox)

INTERVENTIONS:
Drug: CAT-8015 (Moxetumomab Pasudotox) — Participants received intravenous infusion of 5 mcg/kg moxetumomab pasudotox (CAT-8015) without concomitant corticosteroid administration every other day (QoD) in a 21-day cycle for a total of 6 doses per cycle.
  Arms: 5 microgram per kilogram (mcg/kg)
Drug: CAT-8015 (Moxetumomab Pasudotox) — Participants received intravenous infusion of 10 mcg/kg moxetumomab pasudotox (CAT-8015) without concomitant corticosteroid administration every other day (QoD) in a 21-day cycle for a total of 6 doses per cycle.
  Arms: 10 microgram per kilogram (mcg/kg)
Drug: CAT-8015 (Moxetumomab Pasudotox) — Participants received intravenous infusion of 20 mcg/kg moxetumomab pasudotox (CAT-8015) without concomitant corticosteroid administration every other day (QoD) in a 21-day cycle for a total of 6 doses per cycle.
  Arms: 20 microgram per kilogram (mcg/kg): Schema A
Drug: CAT-8015 (Moxetumomab Pasudotox) — Participants received intravenous infusion of 20 mcg/kg moxetumomab pasudotox (CAT-8015) with concomitant corticosteroid administration every other day (QoD) in a 21-day cycle for a total of 6 doses per cycle.
  Arms: 20 microgram per kilogram (mcg/kg): Schema B
Drug: CAT-8015 (Moxetumomab Pasudotox) — Participants received intravenous infusion of 30 mcg/kg moxetumomab pasudotox (CAT-8015) without concomitant corticosteroid administration every other day (QoD) in a 21-day cycle for a total of 6 doses per cycle.
  Arms: 30 microgram per kilogram (mcg/kg): Schema A
Drug: CAT-8015 (Moxetumomab Pasudotox) — Participants received intravenous infusion of 30 mcg/kg moxetumomab pasudotox (CAT-8015) with concomitant corticosteroid administration every other day (QoD) in a 21-day cycle for a total of 6 doses per cycle.
  Arms: 30 microgram per kilogram (mcg/kg): Schema B
Drug: CAT-8015 (Moxetumomab Pasudotox) — Participants received intravenous infusion of 40 mcg/kg moxetumomab pasudotox (CAT-8015) with concomitant corticosteroid administration every other day (QoD) in a 21-day cycle for a total of 6 doses per cycle.
  Arms: 40 microgram per kilogram (mcg/kg): Schema B
Drug: CAT-8015 (Moxetumomab Pasudotox) — Participants received intravenous infusion of 32 mcg/kg moxetumomab pasudotox (CAT-8015) of process 3 material every other day (QoD) in a 21-day cycle for a total of 10 doses per cycle.
  Arms: 32 microgram per kilogram (mcg/kg): Schema C
Drug: CAT-8015 (Moxetumomab Pasudotox) — Participants received intravenous infusion of 50 mcg/kg moxetumomab pasudotox (CAT-8015) without concomitant corticosteroid administration every other day (QoD) in a 21-day cycle for a total of 6 doses per cycle.
  Arms: 50 microgram per kilogram (mcg/kg): Schema B
Drug: CAT-8015 (Moxetumomab Pasudotox) — Participants received intravenous infusion of 50 mcg/kg moxetumomab pasudotox (CAT-8015) continuous every other day (QoD) in a 21-day cycle for a total of 10 doses per cycle.
  Arms: 50 microgram per kilogram (mcg/kg): Schema C

SUMMARY:
A dose-escalation study to estimate maximum cummulative dose (MTCD) of CAT-8015 that can be safely administered to a participant.

DETAILED DESCRIPTION:
A Phase 1, Multicenter, Dose Escalation Study of CAT-8015 in Children, Adolescents and Young Adults with Refractory CD22+ Acute Lymphoblastic Leukemia (ALL) or Non-Hodgkin Lymphoma (NHL) to estimate the maximum tolerated cummulative dose (MTCD), defined as the highest dose and number of doses that can be safely administered to a participant, and to establish a safe dose, based on the MTCD, for subsequent clinical testing.

ELIGIBILITY:
Inclusion Criteria:

- Histologically confirmed diagnosis of acute lymphoblastic leukemia (ALL) or non-Hodgkin's lymphoma (NHL) including lymphoblastic lymphoma, Burkitt's lymphoma, and large cell lymphoma; - Measurable or evaluable disease. - Evidence of CD22-positive malignancy by one of the following criteria: - greater than or equal to (>=) 30 % of malignant cells from a disease site cluster of differentiation 22+ (CD22+) by fluorescence-activated cell sorter (FACS) analysis or; ≥ 15 % of malignant cells from a disease site CD22+ by immunohistochemistry (IHC). Stage of disease: - Participants must have relapsed or refractory disease and have received at least one standard chemotherapy and one salvage regimen or allogeneic stem cell transplant; - Relapse after prior autologous or allogeneic HSCT is allowed. In the event of relapse after prior allogeneic HSCT, the participant must be at least 100 days post-transplant and have no evidence of ongoing active graft-vs-host disease; - Recovered from the acute toxic effects of all prior therapy before entry. Performance status: - Participants greater than or equal to (>=) 12 years of age: Eastern Cooperative Oncology Group (ECOG) score of 0, 1, 2, or 3; - Participants < 12 years of age: Lansky scale >= 50%; - Participants who are unable to walk because of paralysis, but who are up in a wheel chair will be considered ambulatory for the purpose of calculating the performance score. Participants with the following central nervous system (CNS) status, are eligible only in the absence of neurologic symptoms suggestive of CNS leukemia, such as cranial nerve palsy. - Female and male participants with childbearing potential and their sexual partners must agree to use an approved method of contraception during the study.

Exclusion Criteria:

- Participants meeting any of the following criteria are not eligible for participation in the study: - Isolated testicular or CNS ALL; Hepatic function: - Inadequate liver function defined as total bilirubin > 2 × upper limit of normal (ULN) (except in the case of participants with documented Gilbert's disease > 5 × ULN) or transaminases (ALT and aspartate aminotransferase [AST]) > 5 × ULN based on age- and laboratory-specific normal ranges; Renal function: - With greater than age-adjusted normal serum creatinine (see Table below) and a creatinine clearance > 60 millilitre per minute mL/min/1.73 m2. - Age(Years)- Maximum Serum Creatinine (mg/dl)[≤5,0.8] [5 < age less than or equal to 10,1.0] [10 < age less than or equal to 15,1.2 [> 15, 1.5] Hematologic function: - For non-leukemic subjects only, absolute neutrophil count (ANC) < 1000/cmm, or platelet count < 50,000/cmm, if these cytopenias are not judged by the investigator to be due to underlying disease (ie potentially reversible with anti-neoplastic therapy); - Participants with CNS 3 disease; - Hyperleukocytosis (≥ 50,000 blasts/µL) or rapidly progressive disease (PD) that in the estimation of the investigator and sponsor would compromise ability to complete study therapy; - Prior treatment with CAT-3888 (BL22) or any pseudomonas-exotoxin-containing compound; - HIV positive serology (due to increased risk of severe infection and unknown interaction of CAT-8015 with antiretroviral drugs); - Active hepatitis B or C infection.

Ages: 6 Months to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 57 (Actual)
Dates: Start 2008-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medimmune LLC Medimmune LLC, Study Director — MedImmune LLC
Locations (5):
- United States (4):
  - Research Site, Los Angeles, California
  - Research Site, Bethesda, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Memphis, Tennessee
- Research Site, Toronto, Ontario, Canada

REFERENCES:
- [Result] Wayne AS, Shah NN, Bhojwani D, Silverman LB, Whitlock JA, Stetler-Stevenson M, et al. Pediatric phase 1 trial of moxetumomab pasudotox: activity in chemotherapy refractory acute lymphoblastic leukemia (ALL) . http://cancerres.aacrjournals.org/content/74/19_Supplement/CT230.short
- [Derived] Wayne AS, Shah NN, Bhojwani D, Silverman LB, Whitlock JA, Stetler-Stevenson M, Sun W, Liang M, Yang J, Kreitman RJ, Lanasa MC, Pastan I. Phase 1 study of the anti-CD22 immunotoxin moxetumomab pasudotox for childhood acute lymphoblastic leukemia. Blood. 2017 Oct 5;130(14):1620-1627. doi: 10.1182/blood-2017-02-749101. Epub 2017 Aug 9. PMID 28983018

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 57 participants were enrolled of which 55 participants received treatment.
Period: Overall Study
Arm/Group | 5 Microgram Per Kilogram (mcg/kg) | 10 Microgram Per Kilogram (mcg/kg) | 20 Microgram Per Kilogram (mcg/kg): Schema A | 20 Microgram Per Kilogram (mcg/kg): Schema B | 30 Microgram Per Kilogram (mcg/kg): Schema A | 30 Microgram Per Kilogram (mcg/kg): Schema B | 40 Microgram Per Kilogram (mcg/kg): Schema B | 32 Microgram Per Kilogram (mcg/kg): Schema C | 50 Microgram Per Kilogram (mcg/kg): Schema B | 50 Microgram Per Kilogram (mcg/kg): Schema C
Started | 1 | 1 | 1 | 4 | 4 | 5 | 8 | 11 | 6 | 14
Completed | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Not Completed | 1 | 1 | 1 | 4 | 4 | 4 | 8 | 11 | 6 | 13
Not completed — Disease progression | 1 | 0 | 0 | 1 | 0 | 2 | 4 | 3 | 5 | 3
Not completed — Death | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 1 | 4
Not completed — Investigator Discretion | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 0
Not completed — Other | 0 | 1 | 1 | 2 | 4 | 0 | 3 | 2 | 0 | 6

BASELINE CHARACTERISTICS:
Population: Safety Population includes all participants who received any treatment of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | 5 Microgram Per Kilogram (mcg/kg) | 10 Microgram Per Kilogram (mcg/kg) | 20 Microgram Per Kilogram (mcg/kg): Schema A | 20 Microgram Per Kilogram (mcg/kg): Schema B | 30 Microgram Per Kilogram (mcg/kg): Schema A | 30 Microgram Per Kilogram (mcg/kg): Schema B | 40 Microgram Per Kilogram (mcg/kg): Schema B | 32 Microgram Per Kilogram (mcg/kg): Schema C | 50 Microgram Per Kilogram (mcg/kg): Schema B | 50 Microgram Per Kilogram (mcg/kg): Schema C | Total
Number analyzed (Participants) | 1 | 1 | 1 | 4 | 4 | 5 | 8 | 11 | 6 | 14 | 55
Age, Continuous [Mean (Standard Deviation); unit: Years] | 17 (NA) — Standard Deviation is not evaluable for single participant. | 8 (NA) — Standard Deviation is not evaluable for single participant. | 17 (NA) — Standard Deviation is not evaluable for single participant. | 12.8 (6.8) | 9 (2.7) | 14 (4.7) | 8.6 (5.3) | 13.8 (6.3) | 12.8 (8.3) | 14.3 (5.5) | 12.7 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 0 | 3 | 0 | 0 | 3 | 6 | 2 | 6 | 21
  Male | 0 | 1 | 1 | 1 | 4 | 5 | 5 | 5 | 4 | 8 | 34

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: Adverse events that were suspected of a relationship to moxetumomab pasudotox and were greater than or equal to (>=) Grade 3 in severity were considered DLTs with the following additional criteria or exceptions: Participants with hematologic abnormalities of any grade, Grade 2 allergic reactions of bronchospasm or urticaria, or any Grade ≥ 3 allergic reaction, in the presence of premedication.
Time Frame: Day 1 up to 21 days of Cycle 1 (each cycle duration was of 21 days)
Population: Evaluable Population for DLT included all participants who received any treatment of moxetumomab pasudotox (CAT-8015) and completed the DLT period without a DLT, or did not complete the DLT period due to a DLT. Here, "N" is number of participants evaluated for this outcome measure.
Measure: Number; unit: participants
Arm/Group | 10 Microgram Per Kilogram (mcg/kg) | 20 Microgram Per Kilogram (mcg/kg): Schema A | 20 Microgram Per Kilogram (mcg/kg): Schema B | 30 Microgram Per Kilogram (mcg/kg): Schema A | 30 Microgram Per Kilogram (mcg/kg): Schema B | 40 Microgram Per Kilogram (mcg/kg): Schema B | 32 Microgram Per Kilogram (mcg/kg): Schema C | 50 Microgram Per Kilogram (mcg/kg): Schema B | 50 Microgram Per Kilogram (mcg/kg): Schema C
Number analyzed (Participants) | 1 | 1 | 3 | 4 | 3 | 7 | 7 | 3 | 11
participants | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 1

2. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) was any untoward medical occurrence attributed to study drug in a participant who received investigational product. A serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent were events between administration of investigational product and 30 days after the last dose of study drug that were absent before treatment or that worsened relative to pre-treatment state.
Time Frame: From start of study drug administration until 30 days after the last dose of study drug
Population: Safety Population included all participants who received any treatment of study drug.
Measure: Number; unit: Participants
Arm/Group | 5 Microgram Per Kilogram (mcg/kg) | 10 Microgram Per Kilogram (mcg/kg) | 20 Microgram Per Kilogram (mcg/kg): Schema A | 20 Microgram Per Kilogram (mcg/kg): Schema B | 30 Microgram Per Kilogram (mcg/kg): Schema A | 30 Microgram Per Kilogram (mcg/kg): Schema B | 40 Microgram Per Kilogram (mcg/kg): Schema B | 32 Microgram Per Kilogram (mcg/kg): Schema C | 50 Microgram Per Kilogram (mcg/kg): Schema B | 50 Microgram Per Kilogram (mcg/kg): Schema C
Number analyzed (Participants) | 1 | 1 | 1 | 4 | 4 | 5 | 8 | 11 | 6 | 14
Participants
  TEAEs | 1 | 1 | 1 | 4 | 4 | 5 | 8 | 11 | 6 | 14
  TESAEs | 1 | 1 | 1 | 4 | 3 | 2 | 5 | 7 | 4 | 9

3. Primary Outcome: Number of Participants With Vital Signs Abnormalities Recorded as Treatment-Emergent Adverse Events (TEAEs)
Description: Vital signs included parameters as heart rate, blood pressure, temperature, weight, pulse oximetry and respiratory rate. TEAEs were events present at baseline that worsened in intensity after administration of study drug or events absent at baseline that emerged after administration of study drug, for the period extending to 30 days after the last dose of study drug.
Time Frame: From start of study drug administration until 30 days after the last dose of study drug
Population: Safety Population included all participants who received any treatment of study drug.
Measure: Number; unit: Participants
Arm/Group | 5 Microgram Per Kilogram (mcg/kg) | 10 Microgram Per Kilogram (mcg/kg) | 20 Microgram Per Kilogram (mcg/kg): Schema A | 20 Microgram Per Kilogram (mcg/kg): Schema B | 30 Microgram Per Kilogram (mcg/kg): Schema A | 30 Microgram Per Kilogram (mcg/kg): Schema B | 40 Microgram Per Kilogram (mcg/kg): Schema B | 32 Microgram Per Kilogram (mcg/kg): Schema C | 50 Microgram Per Kilogram (mcg/kg): Schema B | 50 Microgram Per Kilogram (mcg/kg): Schema C
Number analyzed (Participants) | 1 | 1 | 1 | 4 | 4 | 5 | 8 | 11 | 6 | 14
Participants
  Tachycardia | 0 | 0 | 0 | 2 | 3 | 3 | 2 | 2 | 0 | 3
  Arrhythmia | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Bradycardia | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1
  Sinus bradycardia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Sinus tachycardia | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Pyrexia | 1 | 0 | 0 | 2 | 4 | 2 | 2 | 2 | 2 | 7
  Dyspnoea | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 4
  Respiratory distress | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2
  Tachypnoea | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0
  Hypertension | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 3 | 1 | 5
  Hypotension | 0 | 1 | 0 | 0 | 1 | 2 | 2 | 2 | 1 | 1

4. Primary Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities Recorded as Treatment-Emergent Adverse Events (TEAEs)
Description: An abnormal laboratory finding which required an action or intervention by the investigator, or a finding judged by the investigator to represent a change beyond the range of normal physiologic fluctuation were reported as an adverse event. Treatment-emergent were events between first dose of study drug and 30 days after the last dose that were absent before treatment or that worsened relative to pretreatment state. Number of participants with grade 3 or higher treatment-emergent adverse events (5% cut off) for laboratory abnormalities were reported as clinically relevant laboratory changes.
Time Frame: From start of study drug administration up to 30 days after the last dose of study drug
Population: Safety population included all participants who received any treatment of study drug.
Measure: Number; unit: Participants
Arm/Group | 5 Microgram Per Kilogram (mcg/kg) | 10 Microgram Per Kilogram (mcg/kg) | 20 Microgram Per Kilogram (mcg/kg): Schema A | 20 Microgram Per Kilogram (mcg/kg): Schema B | 30 Microgram Per Kilogram (mcg/kg): Schema A | 30 Microgram Per Kilogram (mcg/kg): Schema B | 40 Microgram Per Kilogram (mcg/kg): Schema B | 32 Microgram Per Kilogram (mcg/kg): Schema C | 50 Microgram Per Kilogram (mcg/kg): Schema B | 50 Microgram Per Kilogram (mcg/kg): Schema C
Number analyzed (Participants) | 1 | 1 | 1 | 4 | 4 | 5 | 8 | 11 | 6 | 14
Participants
  Febrile neutropenia | 0 | 1 | 1 | 1 | 2 | 1 | 3 | 5 | 0 | 1
  Anemia | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3
  Leukopenia | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 1
  Lymphopenia | 0 | 1 | 1 | 0 | 0 | 1 | 3 | 0 | 0 | 1
  Neutropenia | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Thrombocytopenia | 0 | 1 | 1 | 0 | 0 | 1 | 3 | 1 | 0 | 1

5. Primary Outcome: Treatment-Emergent Adverse Events (TEAEs) Related to Chemistry Abnormalities Occurring in Greater Than (>) 5 Percent of Participants
Description: An abnormal chemistry finding which required an action or intervention by the investigator, or a finding judged by the investigator to represent a change beyond the range of normal physiologic fluctuation were reported as an adverse event. Treatment-emergent were events between first dose of study drug and 30 days after the last dose that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: From start of study drug administration up to 30 days after the last dose of study drug
Population: Safety population included all participants who received any treatment of study drug.
Measure: Number; unit: Participants
Arm/Group | 5 Microgram Per Kilogram (mcg/kg) | 10 Microgram Per Kilogram (mcg/kg) | 20 Microgram Per Kilogram (mcg/kg): Schema A | 20 Microgram Per Kilogram (mcg/kg): Schema B | 30 Microgram Per Kilogram (mcg/kg): Schema A | 30 Microgram Per Kilogram (mcg/kg): Schema B | 40 Microgram Per Kilogram (mcg/kg): Schema B | 32 Microgram Per Kilogram (mcg/kg): Schema C | 50 Microgram Per Kilogram (mcg/kg): Schema B | 50 Microgram Per Kilogram (mcg/kg): Schema C
Number analyzed (Participants) | 1 | 1 | 1 | 4 | 4 | 5 | 8 | 11 | 6 | 14
Participants
  Alanine aminotransferase increased | 0 | 1 | 0 | 2 | 0 | 4 | 2 | 2 | 2 | 3
  Aspartate aminotransferase increased | 1 | 1 | 1 | 0 | 1 | 3 | 5 | 2 | 4 | 2
  Blood creatinine increased | 1 | 0 | 1 | 0 | 2 | 0 | 1 | 1 | 1 | 6
  Blood lactate dehydrogenase increased | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 3 | 0
  Blood urea increased | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 2 | 0
  Hyperglycaemia | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 1 | 2
  Hyperphosphataemia | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
  Hypoalbuminaemia | 0 | 1 | 1 | 0 | 3 | 0 | 1 | 2 | 1 | 2
  Hypocalcaemia | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1
  Hypokalaemia | 1 | 1 | 1 | 1 | 0 | 2 | 4 | 1 | 0 | 1
  Hypomagnesaemia | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
  Hyponatraemia | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 2 | 1
  Hypophosphataemia | 1 | 1 | 0 | 0 | 0 | 0 | 4 | 0 | 1 | 1

6. Primary Outcome: Number of Participants With Abnormalities in Ophthalmologic Examination at End of Treatment That Were Not Present at Baseline
Description: Ophthalmologic examination included evaluation of retinal, corneal and lens abnormalities at baseline and end of treatment that were not present at screening. Participants who experienced abnormalitities during ophthalmologic examination recorded and reported.
Time Frame: Baseline and end of treatment (up to 1 year after the last participants begins study drug treatment)
Population: Safety population included all participants who received any treatment of study drug.
Measure: Number; unit: Participants
Arm/Group | 5 Microgram Per Kilogram (mcg/kg) | 10 Microgram Per Kilogram (mcg/kg) | 20 Microgram Per Kilogram (mcg/kg): Schema A | 20 Microgram Per Kilogram (mcg/kg): Schema B | 30 Microgram Per Kilogram (mcg/kg): Schema A | 30 Microgram Per Kilogram (mcg/kg): Schema B | 40 Microgram Per Kilogram (mcg/kg): Schema B | 32 Microgram Per Kilogram (mcg/kg): Schema C | 50 Microgram Per Kilogram (mcg/kg): Schema B | 50 Microgram Per Kilogram (mcg/kg): Schema C
Number analyzed (Participants) | 1 | 1 | 1 | 4 | 4 | 5 | 8 | 11 | 6 | 14
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

7. Primary Outcome: Number of Participants With Change From Baseline in Normal Sinus Rhythm Findings in ECG
Description: Number of participants with abnormal ECG changes (compared with baseline) as assessed by study cardiologist
Time Frame: Baseline and end of treatment (up to 1 year after the last participant begins study drug treatment)
Population: Safety population included all participants who received any treatment of study drug.
Measure: Number; unit: participants
Arm/Group | 5 Microgram Per Kilogram (mcg/kg) | 10 Microgram Per Kilogram (mcg/kg) | 20 Microgram Per Kilogram (mcg/kg): Schema A | 20 Microgram Per Kilogram (mcg/kg): Schema B | 30 Microgram Per Kilogram (mcg/kg): Schema A | 30 Microgram Per Kilogram (mcg/kg): Schema B | 40 Microgram Per Kilogram (mcg/kg): Schema B | 32 Microgram Per Kilogram (mcg/kg): Schema C | 50 Microgram Per Kilogram (mcg/kg): Schema B | 50 Microgram Per Kilogram (mcg/kg): Schema C
Number analyzed (Participants) | 1 | 1 | 1 | 4 | 4 | 4 | 7 | 7 | 6 | 12
participants | 0 [0.2 to 0.2] | 0 [3.6 to 3.6] | 0 [1.7 to 1.7] | 0 [0.6 to 31.3] | 0 [0.7 to 1.4] | 0 [1.6 to 9.0] | 0 [1.8 to 42.0] | 0 [1.7 to 13.7] | 0 [0.9 to 7.9] | 0 [1.9 to 26.1]

8. Primary Outcome: Change From Baseline to End of Treatment in Clinical Findings in Electrocardiogram (ECG) QT, QTC Interval and Ventricular Rate
Description: The 12-lead ECG data were summarized and evaluated for the following parameters: ,QT, QTC intervals and ventricular rate. Change from baseline in these parameters were reported.
Time Frame: Baseline and end of treatment (up to 1 year after the last participants begins study drug treatment)
Population: Safety population included all participants who received any treatment of study drug.
Measure: Mean (Standard Deviation); unit: milli seconds (msec)
Arm/Group | 5 Microgram Per Kilogram (mcg/kg) | 10 Microgram Per Kilogram (mcg/kg) | 20 Microgram Per Kilogram (mcg/kg): Schema A | 20 Microgram Per Kilogram (mcg/kg): Schema B | 30 Microgram Per Kilogram (mcg/kg): Schema A | 30 Microgram Per Kilogram (mcg/kg): Schema B | 40 Microgram Per Kilogram (mcg/kg): Schema B | 32 Microgram Per Kilogram (mcg/kg): Schema C | 50 Microgram Per Kilogram (mcg/kg): Schema B | 50 Microgram Per Kilogram (mcg/kg): Schema C
Number analyzed (Participants) | 1 | 1 | 1 | 4 | 4 | 5 | 8 | 11 | 6 | 14
milli seconds (msec)
  QT interval | -107 (NA) — Only 1 subject analyzed at baseline and end of treatment so SD is not applicable | NA (NA) — No data available at end of treatment so change from baseline to end of treatment cannot be calculated | NA (NA) — No data available at end of treatment so change from baseline to end of treatment cannot be calculated | NA (NA) — No data available at end of treatment so change from baseline to end of treatment cannot be calculated | -52.0 (NA) — Of the 4 subjects with data, only 1 subject had analyzable data at baseline and end of treatment so SD is not applicable | NA (NA) — No data available at end of treatment so change from baseline to end of treatment cannot be calculated | NA (NA) — No data available at end of treatment so change from baseline to end of treatment cannot be calculated | NA (NA) — No data available at end of treatment so change from baseline to end of treatment cannot be calculated | NA (NA) — No data available at end of treatment so change from baseline to end of treatment cannot be calculated | NA (NA) — No data available at end of treatment so change from baseline to end of treatment cannot be calculated
  QTC interval | 20.0 (NA) — Only 1 subject analyzed at baseline and end of treatment so SD is not applicable | NA (NA) — No data available at end of treatment so change from baseline to end of treatment cannot be calculated | NA (NA) — No data available at end of treatment so change from baseline to end of treatment cannot be calculated | NA (NA) — No data available at end of treatment so change from baseline to end of treatment cannot be calculated | -26.0 (NA) — Of the 4 subjects with data, only 1 subject had analyzable data at baseline and end of treatment so SD is not applicable | NA (NA) — No data available at end of treatment so change from baseline to end of treatment cannot be calculated | NA (NA) — No data available at end of treatment so change from baseline to end of treatment cannot be calculated | NA (NA) — No data available at end of treatment so change from baseline to end of treatment cannot be calculated | NA (NA) — No data available at end of treatment so change from baseline to end of treatment cannot be calculated | NA (NA) — No data available at end of treatment so change from baseline to end of treatment cannot be calculated
  Ventricluar rate | 69.0 (NA) — Only 1 subject analyzed at baseline and end of treatment so SD is not applicable | NA (NA) — No data available at end of treatment so change from baseline to end of treatment cannot be calculated | NA (NA) — No data available at end of treatment so change from baseline to end of treatment cannot be calculated | NA (NA) — No data available at end of treatment so change from baseline to end of treatment cannot be calculated | 29.0 (NA) — Of the 4 subjects with data, only 1 subject had analyzable data at baseline and end of treatment so SD is not applicable | NA (NA) — No data available at end of treatment so change from baseline to end of treatment cannot be calculated | NA (NA) — No data available at end of treatment so change from baseline to end of treatment cannot be calculated | NA (NA) — No data available at end of treatment so change from baseline to end of treatment cannot be calculated | NA (NA) — No data available at end of treatment so change from baseline to end of treatment cannot be calculated | NA (NA) — No data available at end of treatment so change from baseline to end of treatment cannot be calculated

9. Primary Outcome: Best Overall Tumor Response
Description: Antitumor activity was assessed by best overall tumor response.
Time Frame: Baseline and end of treatment (up to 1 year after the last participant begins study drug treatment)
Population: Evaluable Population for Efficacy included all participants who received any treatment of moxetumomab pasudotox and had at least 1 disease assessment after the initiation of moxetumomab pasudotox. Here, "N" is number of participants analyzed for this outcome measure.
Measure: Number; unit: Participants
Arm/Group | 5 Microgram Per Kilogram (mcg/kg) | 10 Microgram Per Kilogram (mcg/kg) | 20 Microgram Per Kilogram (mcg/kg): Schema A | 20 Microgram Per Kilogram (mcg/kg): Schema B | 30 Microgram Per Kilogram (mcg/kg): Schema A | 30 Microgram Per Kilogram (mcg/kg): Schema B | 40 Microgram Per Kilogram (mcg/kg): Schema B | 32 Microgram Per Kilogram (mcg/kg): Schema C | 50 Microgram Per Kilogram (mcg/kg): Schema B | 50 Microgram Per Kilogram (mcg/kg): Schema C
Number analyzed (Participants) | 1 | 1 | 1 | 4 | 4 | 4 | 7 | 7 | 6 | 12
Participants
  Composite complete response | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 2 | 2 | 3
  Complete response | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 2 | 2 | 3
  complete response with incomplete count recovery | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Partial response | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2
  Hematological activity | 0 | 0 | 0 | 2 | 3 | 0 | 3 | 1 | 1 | 2
  Stable disease | 0 | 0 | 1 | 1 | 1 | 1 | 2 | 1 | 0 | 4
  Progressive disease | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 3 | 1

10. Primary Outcome: Objective Response Rate (ORR)
Description: Objective response based on assessment of confirmed composite complete response (CRc) or partial response (PR) according to disease specific criteria [modified criteria for response in acute lymphoblastic leukemia (ALL)].
Time Frame: Baseline until end of treatment (up to 1 year after the last participant begins study drug treatment)
Population: Efficacy population included all participants who received any treatment of study drug and had at least 1 disease assessment after the initiation of study drug. Here, "N" is number of participants analyzed for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | 5 Microgram Per Kilogram (mcg/kg) | 10 Microgram Per Kilogram (mcg/kg) | 20 Microgram Per Kilogram (mcg/kg): Schema A | 20 Microgram Per Kilogram (mcg/kg): Schema B | 30 Microgram Per Kilogram (mcg/kg): Schema A | 30 Microgram Per Kilogram (mcg/kg): Schema B | 40 Microgram Per Kilogram (mcg/kg): Schema B | 32 Microgram Per Kilogram (mcg/kg): Schema C | 50 Microgram Per Kilogram (mcg/kg): Schema B | 50 Microgram Per Kilogram (mcg/kg): Schema C
Number analyzed (Participants) | 1 | 1 | 1 | 4 | 4 | 4 | 7 | 7 | 6 | 12
percentage of participants | 0 | 100 | 0 | 25.0 | 0 | 50.0 | 14.3 | 42.9 | 33.3 | 41.7

11. Primary Outcome: Percentage of Participants With Relapse of Disease
Description: Relapse is defined as progressive disease (PD) following complete response (CR). Rate of relapse was only calculated for the subgroup of participants with complete response.
Time Frame: Baseline until end of treatment (up to 1 year after the last participant begins study drug treatment)
Population: Efficacy population. Here, "N" is number of participants with CR in the respective cohort. Rate of relapse could not be estimated as none of the participants experienced CR in the 5 mcg/kg, 20 mcg/kg (Schema A) and 30 mcg/kg (schema A) cohort of the study.
Measure: Number; unit: percentage of participants
Arm/Group | 5 Microgram Per Kilogram (mcg/kg) | 10 Microgram Per Kilogram (mcg/kg) | 20 Microgram Per Kilogram (mcg/kg): Schema A | 20 Microgram Per Kilogram (mcg/kg): Schema B | 30 Microgram Per Kilogram (mcg/kg): Schema A | 30 Microgram Per Kilogram (mcg/kg): Schema B | 40 Microgram Per Kilogram (mcg/kg): Schema B | 32 Microgram Per Kilogram (mcg/kg): Schema C | 50 Microgram Per Kilogram (mcg/kg): Schema B | 50 Microgram Per Kilogram (mcg/kg): Schema C
Number analyzed (Participants) | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 2 | 3
percentage of participants |  | 0 |  | 100 |  | 0 | 0 | 0 | 50 | 0

12. Primary Outcome: Time to Disease Response
Description: Time to disease response was measured from the start of moxetumomab pasudotox administration to the first documentation of response (CR or PR) and was assessed in participants who achieved objective response.
Time Frame: Baseline and end of treatment (up to 1 year after the last participant begins study drug treatment)
Population: Evaluable Population for Efficacy. Here, "N" is number of participants with objective disease response in the respective cohort. Time to disease response could not be estimated as none of the participants experienced OR in the 5 mcg/kg, 20 mcg/kg (schema A) and 30 mcg/kg (schema A).
Measure: Median (Full Range); unit: months
Arm/Group | 5 Microgram Per Kilogram (mcg/kg) | 10 Microgram Per Kilogram (mcg/kg) | 20 Microgram Per Kilogram (mcg/kg): Schema A | 20 Microgram Per Kilogram (mcg/kg): Schema B | 30 Microgram Per Kilogram (mcg/kg): Schema A | 30 Microgram Per Kilogram (mcg/kg): Schema B | 40 Microgram Per Kilogram (mcg/kg): Schema B | 32 Microgram Per Kilogram (mcg/kg): Schema C | 50 Microgram Per Kilogram (mcg/kg): Schema B | 50 Microgram Per Kilogram (mcg/kg): Schema C
Number analyzed (Participants) | 0 | 1 | 0 | 1 | 0 | 2 | 1 | 3 | 2 | 5
months |  | 0.69 [0.69 to 0.69] |  | 0.49 [0.49 to 0.49] |  | 0.66 [0.59 to 0.72] | 0.49 [0.49 to 0.49] | 0.72 [0.72 to 0.76] | 0.62 [0.59 to 0.66] | 0.66 [0.59 to 0.72]

13. Primary Outcome: Duration of Response (DR)
Description: Duration of response was defined as the duration from the first documentation of objective response to the first documented disease progression.
Time Frame: Baseline and end of treatment (up to 1 year after the last participant begins study drug treatment
Population: Evaluable Population for Efficacy. Here, "N" is number of participants with objective disease response in the respective cohort. DR could not be estimated as none of the participants experienced OR in the 5 mcg/kg, 20 mcg/kg (schema A) and 30 mcg/kg (schema A).
Measure: Median (Full Range); unit: months
Arm/Group | 5 Microgram Per Kilogram (mcg/kg) | 10 Microgram Per Kilogram (mcg/kg) | 20 Microgram Per Kilogram (mcg/kg): Schema A | 20 Microgram Per Kilogram (mcg/kg): Schema B | 30 Microgram Per Kilogram (mcg/kg): Schema A | 30 Microgram Per Kilogram (mcg/kg): Schema B | 40 Microgram Per Kilogram (mcg/kg): Schema B | 32 Microgram Per Kilogram (mcg/kg): Schema C | 50 Microgram Per Kilogram (mcg/kg): Schema B | 50 Microgram Per Kilogram (mcg/kg): Schema C
Number analyzed (Participants) | 0 | 1 | 0 | 1 | 0 | 2 | 1 | 3 | 2 | 5
months |  | NA [1.9 to 1.9] — Median DR was estimated using the Kaplan-Meier survival analysis. Where median DR = NA, it could not be estimated using this method (range is calculated using simple summary statistics) |  | 2.3 [2.3 to 2.3] |  | NA [0.7 to 1.4] — Median DR was estimated using the Kaplan-Meier survival analysis. Where median DR = NA, it could not be estimated using this method (range is calculated using simple summary statistics) | NA [0.8 to 0.8] — Median DR was estimated using the Kaplan-Meier survival analysis. Where median DR = NA, it could not be estimated using this method (range is calculated using simple summary statistics) | NA [0.0 to 0.9] — Median DR was estimated using the Kaplan-Meier survival analysis. Where median DR = NA, it could not be estimated using this method (range is calculated using simple summary statistics) | NA [0.4 to 1.4] — Median DR was estimated using the Kaplan-Meier survival analysis. Where median DR = NA, it could not be estimated using this method (range is calculated using simple summary statistics) | NA [0.0 to 2.0] — Median DR was estimated using the Kaplan-Meier survival analysis. Where median DR = NA, it could not be estimated using this method (range is calculated using simple summary statistics)

14. Primary Outcome: Time to Disease Progression (TDP)
Description: Time to disease progression was measured from the start of treatment with moxetumomab pasudotox until the documentation of disease progression. Number of progressions were reported here.
Time Frame: Baseline and end of treatment (up to 1 year after the last participant begins study drug treatment
Population: as for outcome 9
Measure: Median (Full Range); unit: months
Arm/Group | 5 Microgram Per Kilogram (mcg/kg) | 10 Microgram Per Kilogram (mcg/kg) | 20 Microgram Per Kilogram (mcg/kg): Schema A | 20 Microgram Per Kilogram (mcg/kg): Schema B | 30 Microgram Per Kilogram (mcg/kg): Schema A | 30 Microgram Per Kilogram (mcg/kg): Schema B | 40 Microgram Per Kilogram (mcg/kg): Schema B | 32 Microgram Per Kilogram (mcg/kg): Schema C | 50 Microgram Per Kilogram (mcg/kg): Schema B | 50 Microgram Per Kilogram (mcg/kg): Schema C
Number analyzed (Participants) | 1 | 1 | 1 | 4 | 4 | 4 | 7 | 7 | 6 | 12
months | 0.2 [0.2 to 0.2] | NA [2.6 to 2.6] — Median TDP was estimated using the Kaplan-Meier survival analysis. Where median TDP = NA, it could not be estimated using this method (range is calculated using simple summary statistics) | NA [0.6 to 0.6] — Median TDP was estimated using the Kaplan-Meier survival analysis. Where median TDP = NA, it could not be estimated using this method (range is calculated using simple summary statistics) | 2 [0.5 to 2.8] | NA [0.2 to 1.4] — Median TDP was estimated using the Kaplan-Meier survival analysis. Where median TDP = NA, it could not be estimated using this method (range is calculated using simple summary statistics) | NA [0.5 to 2.2] — Median TDP was estimated using the Kaplan-Meier survival analysis. Where median TDP = NA, it could not be estimated using this method (range is calculated using simple summary statistics) | 1.2 [0.5 to 1.2] | 1.5 [0.5 to 1.6] | 0.8 [0.4 to 2.0] | NA [0.5 to 2.7] — Median TDP was estimated using the Kaplan-Meier survival analysis. Where median TDP = NA, it could not be estimated using this method (range is calculated using simple summary statistics)

15. Primary Outcome: Progression-Free Survival (PFS)
Description: Progression-free survival was measured from the start of treatment with moxetumomab pasudotox until the documentation of disease progression or death due to any cause, whichever occurs first. Number of progressions/deaths were reported here.
Time Frame: Baseline and end of treatment (up to 1 year after the last participant begins study drug treatment)
Population: as for outcome 9
Measure: Median (Full Range); unit: months
Arm/Group | 5 Microgram Per Kilogram (mcg/kg) | 10 Microgram Per Kilogram (mcg/kg) | 20 Microgram Per Kilogram (mcg/kg): Schema A | 20 Microgram Per Kilogram (mcg/kg): Schema B | 30 Microgram Per Kilogram (mcg/kg): Schema A | 30 Microgram Per Kilogram (mcg/kg): Schema B | 40 Microgram Per Kilogram (mcg/kg): Schema B | 32 Microgram Per Kilogram (mcg/kg): Schema C | 50 Microgram Per Kilogram (mcg/kg): Schema B | 50 Microgram Per Kilogram (mcg/kg): Schema C
Number analyzed (Participants) | 1 | 1 | 1 | 4 | 4 | 4 | 7 | 7 | 6 | 12
months | 0.2 [0.2 to 0.2] | 3.6 [3.6 to 3.6] | 1.7 [1.7 to 1.7] | 1.8 [0.6 to 2.8] | NA [0.2 to 1.4] — Median PFS was estimated using the Kaplan-Meier survival analysis. Where median PFS = NA, it could not be estimated using this method (range is calculated using simple summary statistics) | 3.1 [0.5 to 9.0] | 1.2 [0.6 to 14.0] | 1.5 [0.5 to 5.6] | 0.8 [0.4 to 5.9] | 5.8 [0.5 to 17.3]

16. Primary Outcome: Overall Survival (OS)
Description: Overall survival was determined as the time from the start of treatment with Moxetumomab Pasudotox until death. Number of deaths were reported here.
Time Frame: Baseline and end of treatment (up to 1 year after the last participant begins study drug treatment)
Population: as for outcome 9
Measure: Median (Full Range); unit: months
Arm/Group | 5 Microgram Per Kilogram (mcg/kg) | 10 Microgram Per Kilogram (mcg/kg) | 20 Microgram Per Kilogram (mcg/kg): Schema A | 20 Microgram Per Kilogram (mcg/kg): Schema B | 30 Microgram Per Kilogram (mcg/kg): Schema A | 30 Microgram Per Kilogram (mcg/kg): Schema B | 40 Microgram Per Kilogram (mcg/kg): Schema B | 32 Microgram Per Kilogram (mcg/kg): Schema C | 50 Microgram Per Kilogram (mcg/kg): Schema B | 50 Microgram Per Kilogram (mcg/kg): Schema C
Number analyzed (Participants) | 1 | 1 | 1 | 4 | 4 | 4 | 7 | 7 | 6 | 12
months | 0.2 [0.2 to 0.2] | 3.6 [3.6 to 3.6] | 1.7 [1.7 to 1.7] | 2.1 [0.6 to 31.3] | NA [0.7 to 1.4] — Median OS was estimated using the Kaplan-Meier survival analysis. Where median OS = NA, it could not be estimated using this method (range is calculated using simple summary statistics) | 4.6 [1.6 to 9.0] | 9.4 [1.8 to 42.0] | NA [1.7 to 13.7] — Median OS was estimated using the Kaplan-Meier survival analysis. Where median OS = NA, it could not be estimated using this method (range is calculated using simple summary statistics) | 4.1 [0.9 to 7.9] | 12.7 [1.9 to 26.1]

17. Primary Outcome: Maximum Observed Serum Concentration (Cmax) for Moxetumomab Pasudotox
Description: The Cmax is the maximum observed plasma concentration of Moxetumomab Pasudotox.
Time Frame: Cycles 1, 2 and every 4th cycle: pre-dose, end of infusion (EOI), 1, 1.5, 2.5, 4 and 8 hours post-dose of Dose 1; pre-dose and end of infusion after Dose 6
Population: Evaluable Population for efficacy included all participants who received any treatment of study drug and had at least 1 disease assessment after the initiation of study drug.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Groups:
- 20 Microgram Per Kilogram (mcg/kg): Participants received intravenous infusion of 20 mcg/kg CAT-8015 with/without concomitant corticosteroid administration every other day (QoD) in a 21-day cycle for a total of 6 doses per cycle.
- 30 Microgram Per Kilogram (mcg/kg): Participants received intravenous infusion of 30 mcg/kg CAT-8015 with/without concomitant corticosteroid administration every other day (QoD) in a 21-day cycle for a total of 6 doses per cycle.
- 50 Microgram Per Kilogram (mcg/kg): Participants received intravenous infusion of 50 mcg/kg CAT-8015 without concomitant corticosteroid administration/continuous every other day (QoD) in a 21-day cycle for a total of 6 doses per cycle.
Arm/Group | 5 Microgram Per Kilogram (mcg/kg) | 10 Microgram Per Kilogram (mcg/kg) | 20 Microgram Per Kilogram (mcg/kg) | 30 Microgram Per Kilogram (mcg/kg) | 32 Microgram Per Kilogram (mcg/kg): Schema C | 40 Microgram Per Kilogram (mcg/kg): Schema B | 50 Microgram Per Kilogram (mcg/kg)
Number analyzed (Participants) | 1 | 1 | 5 | 9 | 10 | 6 | 20
nanogram per milliliter (ng/mL) | NA (NA) — Cmax below lower limit of quantification | 126 (NA) — Standard deviation was not evaluable since only 1 participant was evaluated. | 274 (135) | 446 (126) | 446 (156) | 555 (196) | 755 (188)

18. Primary Outcome: Area Under the Serum Concentration Time Curve From Time Zero to Infinity (AUC [0 to Infinity]) for Moxetumomab Pasudotox
Description: The AUC (0 to infinity) is the area under the plasma concentration-time curve from time zero to infinity hours.
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: hour*nanogram per milliliter (h.ng/mL)
Arm/Group | 5 Microgram Per Kilogram (mcg/kg) | 10 Microgram Per Kilogram (mcg/kg) | 20 Microgram Per Kilogram (mcg/kg) | 30 Microgram Per Kilogram (mcg/kg) | 32 Microgram Per Kilogram (mcg/kg): Schema C | 40 Microgram Per Kilogram (mcg/kg): Schema B | 50 Microgram Per Kilogram (mcg/kg)
Number analyzed (Participants) | 1 | 1 | 3 | 8 | 10 | 5 | 20
hour*nanogram per milliliter (h.ng/mL) | NA (NA) — AUC cannot be estimated due to insufficient samples from subject to be able to calculate AUC | NA (NA) — AUC cannot be estimated due to insufficient samples from subject to be able to calculate AUC | 744 (514) | 1060 (508) | 844 (385) | 1320 (554) | 1690 (689)

19. Primary Outcome: Systemic Clearance (CL) for Moxetumomab Pasudotox
Description: The CL is a quantitative measure of the rate at which a drug substance is removed from the body. The total systemic clearance after intravenous dose was estimated by dividing the total administered dose by the plasma area under the plasma concentration-time curve from time zone to infinite time (AUC[0-infinity]).
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: milliliter per hour per kilogram
Arm/Group | 5 Microgram Per Kilogram (mcg/kg) | 10 Microgram Per Kilogram (mcg/kg) | 20 Microgram Per Kilogram (mcg/kg) | 30 Microgram Per Kilogram (mcg/kg) | 32 Microgram Per Kilogram (mcg/kg): Schema C | 40 Microgram Per Kilogram (mcg/kg): Schema B | 50 Microgram Per Kilogram (mcg/kg)
Number analyzed (Participants) | 1 | 1 | 3 | 8 | 10 | 5 | 20
milliliter per hour per kilogram | NA (NA) — CL below lower limit of quantification | NA (NA) — CL below lower limit of quantification | 40.5 (32.3) | 35.4 (18.2) | 47.5 (28.2) | 34.6 (13.2) | 35.3 (14.7)

20. Primary Outcome: Terminal Phase Elimination Half Life (t1/2) for Moxetumomab Pasudotox
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: hour (h)
Arm/Group | 5 Microgram Per Kilogram (mcg/kg) | 10 Microgram Per Kilogram (mcg/kg) | 20 Microgram Per Kilogram (mcg/kg) | 30 Microgram Per Kilogram (mcg/kg) | 32 Microgram Per Kilogram (mcg/kg): Schema C | 40 Microgram Per Kilogram (mcg/kg): Schema B | 50 Microgram Per Kilogram (mcg/kg)
Number analyzed (Participants) | 1 | 1 | 3 | 8 | 10 | 5 | 20
hour (h) | NA (NA) — plasma concentration of moxetumomab pasudotox below the lower limit of quantification therefore t1/2 cannot be estimated | NA (NA) — plasma concentration of moxetumomab pasudotox below the lower limit of quantification therefore t1/2 cannot be estimated | 0.906 (0.545) | 1.32 (0.893) | 0.997 (0.557) | 0.880 (0.522) | 1.38 (0.753)

21. Secondary Outcome: Number of Participants With Positive Anti-Drug Antibody (ADA) and Neutralizing Antibody
Description: Participants tested for immunogenicity to CAT-8015 (moxetumomab pasudotox) prior to enrollment, before each cycle and at end of study. The neutralization assay measures the capacity of participant's plasma (antibodies) to inhibit the binding of moxetumomab pasudotox to its target, cluster of differentiation 22 (CD22), coated onto enzyme linked immunosorbent assay (ELISA) plates. It was used as a direct surrogate for biological activity based on the mechanism of action of this drug. Significant level of neutralizing antibody activity defined as the capacity of test plasma to inhibit greater than (>)50 percentage (%) of the binding of CAT-8015 to CD22 using an ELISA-based method.
Time Frame: Baseline until end of treatment (up to 1 year after the last participant begins study drug treatment)
Population: Safety population included all participants who received any treatment of study drug.
Measure: Number; unit: Participants
Arm/Group | 5 Microgram Per Kilogram (mcg/kg) | 10 Microgram Per Kilogram (mcg/kg) | 20 Microgram Per Kilogram (mcg/kg): Schema A | 20 Microgram Per Kilogram (mcg/kg): Schema B | 30 Microgram Per Kilogram (mcg/kg): Schema A | 30 Microgram Per Kilogram (mcg/kg): Schema B | 40 Microgram Per Kilogram (mcg/kg): Schema B | 32 Microgram Per Kilogram (mcg/kg): Schema C | 50 Microgram Per Kilogram (mcg/kg): Schema B | 50 Microgram Per Kilogram (mcg/kg): Schema C
Number analyzed (Participants) | 1 | 1 | 1 | 4 | 4 | 5 | 8 | 11 | 6 | 14
Participants
  ADA present by screening assay | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 1 | 1
  Neutralizing ADA present by functional assay | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 5 | 0 | 3

22. Secondary Outcome: CD22 Expression Cells in Peripheral Blood by Best Response
Description: Participants malignant cells (peripheral blood) was tested for cluster of differentiation 22 (CD22) expression by fluorescence-activated cell sorter (FACS) analysis.
Time Frame: Baseline until end of treatment (up to 1 year after the last participant begins study drug treatment)
Population: Safety population included all participants who received any treatment of study drug. Here, n = participants evaluable for specified category for each arm, respectively
Measure: Median (Full Range); unit: sites per cell
Arm/Group | 5 Microgram Per Kilogram (mcg/kg) | 10 Microgram Per Kilogram (mcg/kg) | 20 Microgram Per Kilogram (mcg/kg): Schema A | 20 Microgram Per Kilogram (mcg/kg): Schema B | 30 Microgram Per Kilogram (mcg/kg): Schema A | 30 Microgram Per Kilogram (mcg/kg): Schema B | 40 Microgram Per Kilogram (mcg/kg): Schema B | 32 Microgram Per Kilogram (mcg/kg): Schema C | 50 Microgram Per Kilogram (mcg/kg): Schema B | 50 Microgram Per Kilogram (mcg/kg): Schema C
Number analyzed (Participants) | 1 | 1 | 1 | 4 | 4 | 5 | 8 | 11 | 6 | 14
sites per cell
  Composite complete response(n=0,1,0,1,0,1,0,2,2,3) | NA [NA to NA] — No participants were evaluated. | 14519.0 [14519 to 14519] | NA [NA to NA] — No participants were evaluated. | 749.0 [749 to 749] | NA [NA to NA] — No participants were evaluated. | 3058.0 [3058 to 3058] | NA [NA to NA] — No participants were evaluated. | 2772.5 [1650 to 3895] | 5620.0 [3968 to 7272] | 4331.0 [3085 to 10393]
  Complete response (n=0,1,0,1,0,1,0,2,2,3) | NA [NA to NA] — No participants were evaluated. | 14519.0 [14519 to 14519] | NA [NA to NA] — No participants were evaluated. | 749.0 [749 to 749] | NA [NA to NA] — No participants were evaluated. | 3058.0 [3058 to 3058] | NA [NA to NA] — No participants were evaluated. | 2772.5 [1650 to 3895] | 5620.0 [3968 to 7272] | 4331.0 [3085 to 10393]
  Partial response (n=0,0,0,0,0,1,0,1,0,2) | NA [NA to NA] — No participants were evaluated. | NA [NA to NA] — No participants were evaluated. | NA [NA to NA] — No participants were evaluated. | NA [NA to NA] — No participants were evaluated. | NA [NA to NA] — No participants were evaluated. | 2387.0 [2387 to 2387] | NA [NA to NA] — No participants were evaluated. | 4514.0 [4514 to 4514] | NA [NA to NA] — No participants were evaluated. | 2366.0 [2312 to 2420]
  Hematological activity (n=0,0,0,2,3,0,3,1,1,2) | NA [NA to NA] — No participants were evaluated. | NA [NA to NA] — No participants were evaluated. | NA [NA to NA] — No participants were evaluated. | 3533.5 [2214 to 4853] | 2476.0 [1851 to 4821] | NA [NA to NA] — No participants were evaluated. | 1427.0 [1194 to 4391] | 1350.0 [1350 to 1350] | 2642.0 [2642 to 2642] | 2223.5 [1616 to 2831]
  Stable response (n=0,0,1,1,1,1,2,1,0,4) | NA [NA to NA] — No participants were evaluated. | NA [NA to NA] — No participants were evaluated. | 5050.0 [5050 to 5050] | 8083.0 [8083 to 8083] | 2111.0 [2111 to 2111] | 5587.0 [5587 to 5587] | 8513.0 [3045 to 13981] | 2521.0 [2521 to 2521] | NA [NA to NA] — No participants were evaluated. | 3904.0 [1226 to 11435]
  Progressive disease (n=1,0,0,0,0,1,1,2,3,1) | 13210.0 [13210 to 13210] | NA [NA to NA] — No participants were evaluated. | NA [NA to NA] — No participants were evaluated. | NA [NA to NA] — No participants were evaluated. | NA [NA to NA] — No participants were evaluated. | 3705.0 [3705 to 3705] | 1415.0 [1415 to 1415] | 5505.5 [1354 to 9657] | 1643.0 [1387 to 5359] | 3102.0 [3102 to 3102]

23. Secondary Outcome: Number of Participants With Potential Biomarkers of Predicting Capillary Leak Syndrome (CLS)
Description: Potential biomarkers include orthostatic blood pressure, albumin levels, weight change, edema and hypoxia were evaluated.
Time Frame: Baseline and end of treatment (up to 1 year after the last participant begins study drug treatment)
Population: Safety population included all participants who received any treatment of study drug.
Measure: Number; unit: participants
Arm/Group | 5 Microgram Per Kilogram (mcg/kg) | 10 Microgram Per Kilogram (mcg/kg) | 20 Microgram Per Kilogram (mcg/kg): Schema A | 20 Microgram Per Kilogram (mcg/kg): Schema B | 30 Microgram Per Kilogram (mcg/kg): Schema A | 30 Microgram Per Kilogram (mcg/kg): Schema B | 40 Microgram Per Kilogram (mcg/kg): Schema B | 32 Microgram Per Kilogram (mcg/kg): Schema C | 50 Microgram Per Kilogram (mcg/kg): Schema B | 50 Microgram Per Kilogram (mcg/kg): Schema C
Number analyzed (Participants) | 1 | 1 | 1 | 4 | 4 | 5 | 8 | 11 | 6 | 14
participants
  Hypertension; Event; Developed no later than CLS | 0 [NA to NA] | 0 [14519 to 14519] | 0 [NA to NA] | 0 [749 to 749] | 0 [NA to NA] | 0 [3058 to 3058] | 0 [NA to NA] | 0 [1650 to 3895] | 0 [3968 to 7272] | 0 [3085 to 10393]
  Hypertension; Event; Developed after CLS | 0 [NA to NA] | 0 [14519 to 14519] | 0 [NA to NA] | 0 [749 to 749] | 2 [NA to NA] | 0 [3058 to 3058] | 0 [NA to NA] | 0 [1650 to 3895] | 0 [3968 to 7272] | 0 [3085 to 10393]
  Hypertension; Event; No CLS | 0 [NA to NA] | 0 [NA to NA] | 0 [NA to NA] | 0 [NA to NA] | 0 [NA to NA] | 0 [2387 to 2387] | 0 [NA to NA] | 2 [4514 to 4514] | 1 [NA to NA] | 5 [2312 to 2420]
  Hypertension; No Event; No CLS | 1 [NA to NA] | 1 [NA to NA] | 1 [NA to NA] | 4 [2214 to 4853] | 2 [1851 to 4821] | 4 [NA to NA] | 8 [1194 to 4391] | 9 [1350 to 1350] | 5 [2642 to 2642] | 8 [1616 to 2831]
  Hypertension; No Event; CLS | 0 [NA to NA] | 0 [NA to NA] | 0 [5050 to 5050] | 0 [8083 to 8083] | 0 [2111 to 2111] | 1 [5587 to 5587] | 0 [3045 to 13981] | 0 [2521 to 2521] | 0 [NA to NA] | 1 [1226 to 11435]
  Weight change; Event; Developed no later than CLS | 0 [13210 to 13210] | 0 [NA to NA] | 0 [NA to NA] | 0 [NA to NA] | 1 [NA to NA] | 0 [3705 to 3705] | 0 [1415 to 1415] | 0 [1354 to 9657] | 0 [1387 to 5359] | 0 [3102 to 3102]
  Weight change; Event; Developed after CLS | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Weight change; Event; No CLS | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 3 | 0 | 3
  Weight change; No Event; No CLS | 1 | 1 | 1 | 2 | 2 | 3 | 8 | 8 | 6 | 10
  Weight change; No Event; CLS | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
  Change in Albumin; Event; Developed no later CLS | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Change in Albumin; Event; Developed after CLS | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Change in Albumin; Event; No CLS | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Change in Albumin; No Event; No CLS | 1 | 1 | 1 | 4 | 2 | 3 | 8 | 11 | 6 | 13
  Change in Albumin; No Event; CLS | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 1
  Edema; Event; Developed no later than CLS | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Edema; Event; Developed after CLS | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Edema; Event; No CLS | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Edema; No Event; No CLS | 1 | 1 | 1 | 4 | 2 | 4 | 8 | 11 | 6 | 13
  Edema; No Event; CLS | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1
  Hypoxia; Event; Developed no later than CLS | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Hypoxia; Event; Developed after CLS | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
  Hypoxia; Event; No CLS | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 2 | 2 | 1
  Hypoxia; No Event; No CLS | 0 | 1 | 0 | 3 | 2 | 4 | 7 | 9 | 4 | 12
  Hypoxia; No Event; CLS | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: From start of study drug administration up to 30 days after the last dose of study drug
Groups:
- 5 UG/KG SCHEMA A: Participants received intravenous infusion of 5 mcg/kg moxetumomab pasudotox (CAT-8015) without concomitant corticosteroid administration every other day (QoD) in a 21-day cycle for a total of 6 doses per cycle.
- 10 UG/KG SCHEMA A: Participants received intravenous infusion of 10 mcg/kg moxetumomab pasudotox (CAT-8015) without concomitant corticosteroid administration every other day (QoD) in a 21-day cycle for a total of 6 doses per cycle.
- 20 UG/KG SCHEMA A: Participants received intravenous infusion of 20 mcg/kg moxetumomab pasudotox (CAT-8015) without concomitant corticosteroid administration every other day (QoD) in a 21-day cycle for a total of 6 doses per cycle.
- 20 UG/KG SCHEMA B: Participants received intravenous infusion of 20 mcg/kg moxetumomab pasudotox (CAT-8015) with concomitant corticosteroid administration every other day (QoD) in a 21-day cycle for a total of 6 doses per cycle.
- 30 UG/KG SCHEMA A: Participants received intravenous infusion of 30 mcg/kg moxetumomab pasudotox (CAT-8015) without concomitant corticosteroid administration every other day (QoD) in a 21-day cycle for a total of 6 doses per cycle.
- 30 UG/KG SCHEMA B: Participants received intravenous infusion of 30 mcg/kg moxetumomab pasudotox (CAT-8015) with concomitant corticosteroid administration every other day (QoD) in a 21-day cycle for a total of 6 doses per cycle.
- 40 UG/KG SCHEMA B: Participants received intravenous infusion of 40 mcg/kg moxetumomab pasudotox (CAT-8015) with concomitant corticosteroid administration every other day (QoD) in a 21-day cycle for a total of 6 doses per cycle.
- 32 UG/KG SCHEMA C: Participants received intravenous infusion of 32 mcg/kg moxetumomab pasudotox (CAT-8015) of process 3 material every other day (QoD) in a 21-day cycle for a total of 10 doses per cycle.
- 50 UG/KG SCHEMA B: Participants received intravenous infusion of 50 mcg/kg moxetumomab pasudotox (CAT-8015) without concomitant corticosteroid administration every other day (QoD) in a 21-day cycle for a total of 6 doses per cycle.
- 50 UG/KG SCHEMA C: Participants received intravenous infusion of 50 mcg/kg moxetumomab pasudotox (CAT-8015) continuous every other day (QoD) in a 21-day cycle for a total of 10 doses per cycle.
Arm/Group | 5 UG/KG SCHEMA A | 10 UG/KG SCHEMA A | 20 UG/KG SCHEMA A | 20 UG/KG SCHEMA B | 30 UG/KG SCHEMA A | 30 UG/KG SCHEMA B | 40 UG/KG SCHEMA B | 32 UG/KG SCHEMA C | 50 UG/KG SCHEMA B | 50 UG/KG SCHEMA C
Serious Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 1/1 | 4/4 | 3/4 | 2/5 | 5/8 | 7/11 | 4/6 | 9/14
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 1/1 | 4/4 | 4/4 | 5/5 | 8/8 | 11/11 | 6/6 | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5 UG/KG SCHEMA A (N=1) | 10 UG/KG SCHEMA A (N=1) | 20 UG/KG SCHEMA A (N=1) | 20 UG/KG SCHEMA B (N=4) | 30 UG/KG SCHEMA A (N=4) | 30 UG/KG SCHEMA B (N=5) | 40 UG/KG SCHEMA B (N=8) | 32 UG/KG SCHEMA C (N=11) | 50 UG/KG SCHEMA B (N=6) | 50 UG/KG SCHEMA C (N=14)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 1 (2) | 1 (1) | 0 (0) | 1 (2) | 2 (3) | 1 (2) | 0 (0) | 0 (0)
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Choroidal detachment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Brain death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Multi-organ failure (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Hepatobiliary disease (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Venoocclusive liver disease (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Geotrichum infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Opportunistic infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia fungal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Acute lymphocytic leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Central nervous system haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coma (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemoglobinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Disease progression (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutropenic infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Systemic mycosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Troponin (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Capillary leak syndrome (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Venoocclusive disease (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5 UG/KG SCHEMA A (N=1) | 10 UG/KG SCHEMA A (N=1) | 20 UG/KG SCHEMA A (N=1) | 20 UG/KG SCHEMA B (N=4) | 30 UG/KG SCHEMA A (N=4) | 30 UG/KG SCHEMA B (N=5) | 40 UG/KG SCHEMA B (N=8) | 32 UG/KG SCHEMA C (N=11) | 50 UG/KG SCHEMA B (N=6) | 50 UG/KG SCHEMA C (N=14)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (19) | 1 (12) | 0 (0) | 0 (0) | 0 (0) | 2 (12) | 0 (0) | 0 (0) | 3 (17)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 4 (4) | 0 (0) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 3 (7) | 0 (0) | 0 (0) | 1 (12)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (13) | 1 (4) | 0 (0) | 0 (0) | 1 (4) | 3 (7) | 0 (0) | 0 (0) | 1 (10)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (7) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (7)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (38) | 1 (8) | 0 (0) | 0 (0) | 1 (12) | 3 (24) | 0 (0) | 0 (0) | 1 (15)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 3 (3) | 3 (4) | 2 (2) | 2 (2) | 0 (0) | 3 (4)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (4) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 3 (5) | 4 (4) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (7) | 0 (0) | 4 (7) | 2 (2) | 0 (0) | 5 (6)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (4) | 1 (3) | 1 (1) | 1 (1) | 0 (0) | 2 (5) | 2 (2) | 0 (0) | 3 (4)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 2 (2)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 4 (4) | 1 (2) | 5 (5)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 4 (8) | 2 (10) | 2 (3) | 2 (6) | 3 (8)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 3 (5) | 5 (10) | 2 (2) | 4 (7) | 2 (5)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (5) | 0 (0)
Blood urea increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (4) | 0 (0) | 2 (3) | 0 (0)
Electrocardiogram qt prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (2) | 1 (1) | 1 (3) | 3 (20) | 2 (11) | 2 (3) | 3 (5) | 1 (3) | 8 (17)
Platelet count decreased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 4 (23) | 4 (33) | 3 (25) | 6 (39) | 4 (17) | 7 (37)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 4 (8) | 2 (6) | 2 (4) | 0 (0) | 7 (15) | 3 (4) | 4 (15)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (16) | 2 (10) | 3 (5) | 1 (8) | 4 (8) | 2 (11) | 8 (43)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 3 (5) | 0 (0) | 1 (1) | 2 (13)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (4) | 0 (0) | 3 (7) | 0 (0) | 1 (1) | 2 (2) | 1 (2) | 2 (4)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (6)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (3) | 1 (2) | 1 (3) | 0 (0) | 2 (3) | 4 (5) | 1 (3) | 0 (0) | 1 (4)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 2 (5) | 1 (3) | 4 (6) | 2 (2) | 7 (10)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (7)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 2 (2)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 1 (1) | 2 (2) | 1 (2) | 4 (7)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 1 (1) | 4 (6)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 2 (3) | 2 (5) | 7 (15)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (6)
Blood creatinine increased (Investigations) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (3) | 6 (13)
Haemoglobin decreased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 3 (8) | 4 (11) | 3 (7) | 2 (10) | 4 (9) | 2 (12) | 8 (38)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (5)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 2 (2) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 1 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 1 (1) | 1 (1) | 2 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Haemoglobinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 1 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (3) | 0 (0) | 2 (2) | 1 (1) | 1 (2)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 2 (4) | 1 (1) | 0 (0) | 1 (2) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 5 (9)
Hypotension (Vascular disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 2 (2) | 1 (1) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.